CLINICAL TRIAL: NCT06387771
Title: Evaluation of the Efficacy of Tolcapone as a Genotype-based Targeted Cognitive Enhancer in Schizophrenia, Based on the Polymorphism rs4680
Brief Title: Evaluation of Tolcapone as a Cognitive Enhancer in Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rs4680-tolcapona
Record Dates: First submitted 2015-09-14; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Pharmacogenetics; fMRI
MeSH Terms: conditions — Schizophrenia | interventions — Tolcapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolcapone (Experimental): Tolcapone (Film-coated tablet) 200 mg orally every 8 hours for 7 days
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone — Tolcapone (Film-coated tablet) 200 mg orally every 8 hours for 7 days

SUMMARY:
Objective: To assess the efficacy of tolcapone to improve cognition in schizophrenia, as a genotype-based targeted treatment of cognitive and negative symptoms of schizophrenia considering the polymorphism rs4680.

Methodology: 20 patients with chronic and stabilized schizophrenia (10 patients with genotype Val/Val and 10 patients with genotype Met/Met according to polymorphism rs4680) will receive treatment with tolcapone during 7 days. The cognitive function and clinical status will be evaluated with a neuropsychological battery and appropriate clinical scales before and after treatment. The efficiency of the activation of the prefrontal cortex will be measured using functional magnetic resonance imaging (fMRI) before and after treatment.

Hypothesis: Only patients with genotype Val/Val treated with tolcapone would show a cognitive improvement, a higher efficiency of the activation of the prefrontal cortex and an amelioration of some negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent and express the wish to fulfill all the requirements of the protocol during the study period.
* The patient must be capable of fulfillment of all the requirements of the clinical trial, at the investigator's discretion.
* Patients diagnosed with schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Only chronic patients will be recruited, and they must be clinically compensated in order to consent to participate. The determination of clinical compensation will be conducted according with these criteria: i) outpatients, with absence of hospitalization due to acute psychiatric decompensation in the previous year, and ii) maintained GAF score equal or higher than 60 during the previous month. The recruitment process will include a clinical interview to verify the diagnosis.
* Caucasic ethnicity
* Negative pregnancy test for women of childbearing age.

Exclusion Criteria:

* Severe infections or diseases or hepatic failure (or increased liver enzymes), renal failure or bone marrow failure that advise against participation in the study at the investigator's discretion
* Positive pregnancy test, or breastfeeding women.
* Carriers of pacemaker or any kind of metallic prosthesis incompatible with magnetic resonance imaging.
* History of hypersensitivity to Tasmar® (tolcapone) or to any of its components
* Active (in the last 12 months) substance abuse, or other disease that causes psychiatric symptoms
* Cardiovascular disease and electrocardiogram alterations
* Patients receiving treatment with monoamine oxidase inhibitors during the study or up to 15 days prior to the beginning of the study.
* Patients receiving treatment with a catechol-O-methyltransferase (COMT) inhibitor
* Participation in another clinical trial in the previous 30 days.
* Other circumstances which involve Tasmar® (tolcapone) contraindications: history of Neuroleptic Malignant Syndrome and/or non-traumatic rhabdomyolysis or hyperthermia. Severe dyskinesia. Phaeochromocytoma. Hereditary galactose intolerance. Lapp lactase deficiency or glucose or galactose malabsorption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09-22 (Actual); Primary Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Change from baseline in cognitive test scores at day 8 | Day 8
  Performance in the cognitive tests scores: Dot Pattern Expectancy Task and cognitive tests (including subtests of the MATRICS* battery) (*MATRICS=Measurement and Treatment Research to Improve Cognition in Schizophrenia cognitive battery established by the National Institute of Mental Health) .
Efficacy: Change from baseline in the brain blood-oxygen-level-dependent (BOLD) response at day 8 | Day 8
  Elicited brain activation during functional magnetic resonance neuroimaging (relative degree of activation of different brain regions) measured by BOLD signal.

SECONDARY OUTCOMES:
Efficacy: change from baseline in psychotic symptoms intensity measured by the PANSS scores at day 8 | Day 8
  Change in psychotic symptoms intensity measured by the PANSS symptom scores
Efficacy: negative symptoms intensity: change from baseline in the 16-item Negative Symptom Assessment (NSA-16) scale scores at day 8 | Day 8
  Change in negative symptoms intensity measured by the NSA-16 scale
Efficacy: change from baseline in the intensity of psychotic symptoms measured by the Brief Psychiatric Rating Scale (BPRS) scores at day 8 | Day 8
  Clinical outcome measured by the change in the scores on the BPRS
Efficacy: change from baseline in the clinical global impression measured by the Clinical Global Impression (CGI) scale scores at day 8 | Day 8
  Clinical outcome measured by the change in the scores on the CGI scale
Efficacy: change from baseline in the global assessment of functioning measured by the Global Assessment of Functioning (GAF) scale scores at day 8 | Day 8
  Clinical outcome measured by the change in the scores on the GAF scale
Efficacy: change from baseline in the anxiety symptoms measured by the Hamilton Anxiety Rating Scale (HAM-A) scale scores at day 8 | Day 8
  Clinical outcome measured by the change in the scores on the HAM-A scale
Efficacy: change from baseline in the depressive symptoms measured by the Hamilton Depression Rating Scale (HAM-D) scale scores at day 8 | Day 8
  Clinical outcome measured by the change in the scores on the HAM-D scale
Efficacy: change from baseline in the Clinician-Rated Dimensions of Psychosis Symptom Severity (CRDPSS) scale scores at day 8 | Day 8
  Clinical outcome measured by the change in the scores on the CRDPSS scale
Change from baseline in plasmatic homocysteine (umol/L) | Day 8
  Clinical outcome measured by the change in homocystinemia (umol/L)

OTHER OUTCOMES:
Patient Reported Outcome: change from baseline in the Profile of Mood States (POMS) scores at day 8 | Day 8
  Patient Reported Outcome measured by the change in the POMS scores
Patient Reported Outcome: change from baseline in the mood state Visual Analogue Scale (VAS) scores at day 8 | Day 8
  Patient Reported Outcome measured by the change in the mood state VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Molero, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain